CLINICAL TRIAL: NCT03249337
Title: A Pilot Study For Efficacy And Safety Of Glanatec® Opthalmic Solution 0.4% On Corneal Edema And Endothelial Cell Counts In Subjects With Fuchs Endothelial Dystrophy Undergoing Descemet Stripping Without Endothelial Keratoplasty
Brief Title: Glanatec(R) for Descemet Stripping in Fuch's Endothelial Dystrophy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marian Macsai, MD (Other)
Responsible Party: Sponsor-Investigator, Marian Macsai, MD, Chief Ophthalmology, Endeavor Health
Organization: Endeavor Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH17-320
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Ophthalmic Solutions; K-115

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glanatec(R) 3 times a day (Active Comparator)
  Interventions: Drug: Ripasudil hydrochloride hydrate 0.4% ophthalmic solution
- Glanatec (R) 6 times a day (Active Comparator)
  Interventions: Drug: Ripasudil hydrochloride hydrate 0.4% ophthalmic solution

INTERVENTIONS:
Drug: Ripasudil hydrochloride hydrate 0.4% ophthalmic solution — the ophthalmic solution will be administered three or six per times per day in the eye designated as the "Study Eye" upon study enrollment
  Other Names: Glanatec

SUMMARY:
In brief, the objective of this study is to investigate whether the drug Glanatec ® which is approved in Japan for glaucoma and ocular hypertension, can be used in patients with Fuchs endothelial dystrophy who have had a descemet stripping procedure without endothelial keratoplasty. While some limited data exists as a proof of concept in in vitro or animal studies, and Glanatec® has been successfully used in a recently published case series for this indication, there is insufficient data to show that this drug can be effectively used for corneal cell clearing while maintaining patient safety.

The goal of the study is to provide sufficient proof of concept for the use of this drug in patients with FED whose only treatment alternative is to undergo corneal transplant.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to understand read and sign the informed consent form.

  * Age between 30 and <91 years
  * Ability to understand and follow instructions and study procedures
  * Willingness to comply with all study procedures and be available for the duration of the study
  * Ability to apply eye drop medication and willing to adhere to study medication regimen
  * Diagnosed with Fuchs dystrophy (clinically and on confocal microscopy) by the study investigator.
  * Pseudophakic FED with posterior capsule supported, suture-fixated, or sulcus-supported posterior chamber intraocular lens.
  * Fuchs dystrophy grades 2-4 on the Krachmer grading scale
  * Presence of central guttae deemed by the investigator to be the chief cause of visual symptoms, rather than cataract or corneal stromal edema
  * Clear peripheral cornea with an endothelial cell count >1000 cells/mm2 on specular microscopy
  * Best corrected visual acuity in the study eye is 20/40 or worse at study enrollment
  * The patient is dissatisfied with current vision
  * The patient is otherwise to be offered a corneal graft
  * For females with reproductive potential, willingness to use highly effective contraception (e.g., hormonal contraception, barrier contraception, intrauterine device, or abstinence).
  * Indication for surgery may include cataract extraction and posterior chamber intraocular lens implantation

Exclusion Criteria:

* • Uncontrolled glaucoma (IOP >25 mmHg)

  * Presence of secondary corneal pathology such as infective or autoimmune keratitis
  * Advanced corneal stromal edema defined as the presence of haze, bullae, or DM folds on slit-lamp biomicroscopy
  * History of herpes simplex virus or cytomegalovirus keratitis
  * Prior endothelial keratoplasty
  * Aphakic in study eye.
  * Allergy to any component of the Ripasudil hydrochloride hydrate 0.4% that will be used in the course of the study
  * For women of child-bearing potential: Pregnant or lactating, or planning to become pregnant within the next 6 months.
  * Any other ocular condition that, in the opinion of the investigator, may preclude the subject from study participation.

Ages: 18 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Corneal Clearing | 12 months
  The first primary aim of this study is to examine whether Glanatec® administered three or six times daily significantly increases corneal clearing at 12 months versus baseline in patients with Fuchs endothelial dystrophy (FED) undergoing Descemet stripping
pachymetry measurement | 12 months
  The second primary aim of this study is to examine whether Glanatec® administered three or six times daily significantly reduces the pachymetry measurement at 12 months versus baseline in patients with Fuchs endothelial dystrophy (FED) undergoing Descemet stripping.

SECONDARY OUTCOMES:
Visual Acuity | 12 months
  The secondary aim of this study is to examine whether Glanatec® administered three or six times daily affects best corrected visual acuity at 12 months (measured by Snellen lines) as compared to baseline, patients with Fuchs endothelial dystrophy (FED) undergoing Descemet stripping.

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Glenview, Illinois, United States

IPD SHARING:
Plan to Share IPD: No